CLINICAL TRIAL: NCT05913791
Title: Impact of Nutrients-fortified Egg Consumption on Eczema Condition in Individuals With Eczema
Brief Title: Nutrients-fortified Egg Consumption on Eczema Condition in Individuals With Eczema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Ministry of Education, Singapore (Other Government)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: S17
Record Dates: First submitted 2023-03-31; First posted 2023-06-22 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Eczema, Atopic; Inflammation; Skin; Eczema; Hypersensitivity
Keywords: Egg; Vitamin D; Vitamin E; Antioxidant; Eczema; Omega-3 long chain polyunsaturated fatty acids
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Eczema; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrients-fortified egg (Experimental): Each subject will be provided with 2 nutrients-fortified eggs from N&N Agriculture Pte Ltd to consume daily for 12 weeks. They will be instructed to consume the eggs for breakfast with the following preparation methods: hard-boiling, half-boiling and steaming. Subjects are to continue their usual diet.
  Interventions: Dietary Supplement: Nutrients-fortified egg
- Regular egg (Placebo Comparator): Each subject will be provided with 2 regular eggs to consume daily for 12 weeks. They will be instructed to consume the eggs for breakfast with the following preparation methods: hard-boiling, half-boiling and steaming. Subjects are to continue their usual diet.
  Interventions: Other: Regular egg

INTERVENTIONS:
Dietary Supplement: Nutrients-fortified egg — Consumption of 2 cooked nutrients fortified eggs (half-boiled, hard-boiled, or steamed)
  Arms: Nutrients-fortified egg
Other: Regular egg — Consumption of 2 regular eggs, prepared in the same manner as nutrients-fortified egg, which serves as a placebo comparison.
  Arms: Regular egg

SUMMARY:
The study aims to assess the effects of daily consumption of nutrients-fortified eggs on eczema condition in individuals with eczema.

It is hypothesised that daily consumption of nutrients-fortified egg, which is rich in antioxidants, will improve eczema conditions in individuals with eczema as compared to consumption of regular eggs.

DETAILED DESCRIPTION:
Eczema refers to a group of conditions that induces inflammation of the skin. Of which, atopic dermatitis is the most common type. Eczema is common in children, and can continue to adulthood. Eczema is a chronic condition with no known cure.

Anti-inflammatory agents have been shown to protect against atopic dermatitis. Vitamin D, E and polyunsaturated fatty acids are known to confer excellent anti-inflammatory benefits.

This is a double-blinded, randomized, parallel study and all subjects will complete a 12-week study period. The study was designed based on previous research which reported that omega-3 supplementation significantly decreased blood IgE concentration (-29.0 ± 11.1, mean ± SD) compared to placebo supplementation (-7.7 ± 14.6, mean ± SD).

ELIGIBILITY:
Inclusion Criteria:

1. English-literate and able to give informed consent in English
2. Male and female subjects, aged between 21 and 59 inclusive
3. Healthy individuals with no comorbidities or on regular medication
4. BMI between 18.5-25 kg/m2
5. Mild to moderate severity of eczema, which will also be determined using our questionnaires during screening visit

Exclusion Criteria:

1. Significant change in body weight (3 kg or more) in the past 3 months
2. Significant exercise pattern over the past 3 months defined as high-intensity exercise of more than 3 hours per week
3. Known food allergy to eggs
4. Taking dietary supplements which may impact the study results
5. Had been diagnosed or with a history of gastrointestinal disorders e.g. irritable bowel syndrome, constipation, diverticulitis
6. Current smokers
7. Consumes more than 2 alcoholic drinks per day i.e. one drink is defined as either 150ml of wine, 340ml of beer/cider or 45ml of distilled spirit
8. Taking lipid-lowering and blood pressure controlling medications less than 3 years
9. Pregnant or lactating women, or planning to conceive in the next 6 months
10. Unwilling to stop the medication of eczema during the study, either topical creams or oral medications
11. Hierarchical link (professional and familial ties) with the research team members
12. Participating in another clinical study
13. Having blindness in one eye or more, previously diagnosed eye diseases, or have had eye surgery
14. Low quality macular pigment optical density results, determined during screening visit

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in eczema severity using the SCORing Atopic Dermatitis (SCORAD) index | Every 3 weeks (Week 0, Week 3, Week 6, Week 9, Week 12)
  The SCORAD index is a validated composite scoring instrument designed to assess signs and symptoms of atopic dermatitis (AD). Total score ranges from 0 to 103, with higher scores indicating greater severity.
Change in eczema severity using the Eczema Area Severity Index (EASI) | Every 3 weeks (Week 0, Week 3, Week 6, Week 9, Week 12)
  The EASI is a validated objective instrument for assessing signs of AD. Total score ranges from 0 to 72, with higher scores indicating greater severity.
Change in skin quality of life assessment using the Dermatology Life Quality Index (DLQI) | Every 3 weeks (Week 0, Week 3, Week 6, Week 9, Week 12)
  The DLQI is a validated self-reported instrument assessing the self perception of impact of skin diseases on their quality of life over the previous week. Scores range from 0 to 30, with higher scores indicating greater impairment on quality of life.
Change in skin hydration level using corneometer | Every 3 weeks (Week 0, Week 3, Week 6, Week 9, Week 12)
  A corneometer is an electronic device used to measure hydration on the skin surface
Change in transepidermal water loss level using tewameter | Every 3 weeks (Week 0, Week 3, Week 6, Week 9, Week 12)
  A tewameter is an electronic device used to measure transepidermal water loss on the skin surface
Change in skin pH level using pH probe | Every 3 weeks (Week 0, Week 3, Week 6, Week 9, Week 12)
  A pH probe is an electronic device used to measure pH levels on the skin surface
Change in skin sebum level using sebumeter | Every 3 weeks (Week 0, Week 3, Week 6, Week 9, Week 12)
  A sebumeter is an electronic device used to measure sebum levels on the skin surface
Change in stratum corneum components via immune dot blot assay | Baseline and Week 12
  Outermost skin surface components will be extracted to conduct dot blot assays to assess changes during intervention period
Change in malondialdehyde level | Every 6 weeks (Week 0, Week 6, Week 12)
  Malondialdehyde concentration in blood samples will be measured
Change in 8-iso-prostaglandin F2α level | Every 6 weeks (Week 0, Week 6, Week 12)
  8-iso-prostaglandin F2α concentration in blood samples will be measured
Change in interleukin-6 level | Every 6 weeks (Week 0, Week 6, Week 12)
  Interleukin-6 concentration in blood samples will be measured
Change in tumor necrosis factor α | Every 6 weeks (Week 0, Week 6, Week 12)
  Tumor necrosis factor α concentration in blood samples will be measured
Change in fasting blood glucose level | Every 6 weeks (Week 0, Week 6, Week 12)
  Fasting glucose concentration in blood samples will be measured
Change in blood triglyceride level | Every 6 weeks (Week 0, Week 6, Week 12)
  Triglyceride concentration in blood samples will be measured
Change in blood total cholesterol level | Every 6 weeks (Week 0, Week 6, Week 12)
  Total cholesterol levels in blood samples will be measured
Change in blood Low-density Lipoprotein-cholesterol (LDL) level | Every 6 weeks (Week 0, Week 6, Week 12)
  LDL concentration in blood samples will be measured
Change in blood High-density Lipoprotein-cholesterol (HDL) level | Every 6 weeks (Week 0, Week 6, Week 12)
  HDL concentration in blood samples will be measured

SECONDARY OUTCOMES:
Change in Blood Carotenoid levels using High Performance Liquid Chromatography (HPLC) | Every 6 weeks (Week 0, Week 6, Week 12)
  Carotenoid concentration in blood samples will be measured
Change in Skin Carotenoid levels using BioPhotonic Scanner | Every 3 weeks (Week 0, Week 3, Week 6, Week 9, Week 12)
  Skin carotenoid levels will be measured from the skin surface
Change in Eye Carotenoid levels using Macular Pigment Scanner | Every 3 weeks (Week 0, Week 3, Week 6, Week 9, Week 12)
  Eye carotenoid levels will be measured using the Macular Pigment Scanner MPSII
Change in Skin Advanced Glycation End-product (AGEs) | Every 3 weeks (Week 0, Week 3, Week 6, Week 9, Week 12)
  Skin AGEs will be quantified using a noninvasive scanner
Change in Blood AGEs | Every 6 weeks (Week 0, Week 6, Week 12)
  Blood AGEs concentration in blood samples will be measured
Change in Eye Visual Function using the NEI VFQ-25 | Every 3 weeks (Week 0, Week 3, Week 6, Week 9, Week 12)
  The National Eye Institute Visual Functioning Questonnaire-25 (NEI VFQ-25) is a self-reported instrument designed to assess visual disability and health-related quality of life. The overall composite score ranges from 0 to 100, with a higher score indicating better visual function and better quality of life.
Change in Visual Acuity using eye chart | Every 3 weeks (Week 0, Week 3, Week 6, Week 9, Week 12)
  Visual acuity is a measure of visual function and it will be assessed by an investigator
Change in Contrast Sensitivity using eye chart | Every 3 weeks (Week 0, Week 3, Week 6, Week 9, Week 12)
  Contrast sensitivity is a measure of visual function and it will be assessed by an investigator
Change in Photostress Recovery Time using eye chart | Every 3 weeks (Week 0, Week 3, Week 6, Week 9, Week 12)
  Photostress recovery assessment is a measure of visual function and it will be assessed by an investigator

CONTACTS AND LOCATIONS:
Overall Officials: Jung Eun Kim, PhD, Principal Investigator — Food Science and technology, Faculty of Science, National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Hard copy documents containing identifiable participant information will be stored in locked storage cabinets accessible only to members of the NUS research group. These locked storage cabinets are located in Kim lab in NUS. This lab is accessible only to Dr Kim Jung Eun, the Principal Investigator, and Dr Kim's research staff. The lab has a dual access security system, with the first entry point being an electronic lock accessible by an NUS-approved key card and the second is a physical lock.
  Electronic copies of the data with identifiable participant information stored electronically in NUS OneDrive. Only members of Dr Kim's lab have access to this secured folder. Access to this OneDrive folder is only granted by Dr Kim.
  All study samples will be de-identified prior to analysis and statistical analyses.

REFERENCES:
- [Background] Ito N, Seki S, Ueda F. The Protective Role of Astaxanthin for UV-Induced Skin Deterioration in Healthy People-A Randomized, Double-Blind, Placebo-Controlled Trial. Nutrients. 2018 Jun 25;10(7):817. doi: 10.3390/nu10070817. PMID 29941810